CLINICAL TRIAL: NCT05578508
Title: A Phase I Study of Bone Marrow Derived Mesenchymal Stem Cells (MSCs) for the Treatment of Medically Refractory Pouchitis
Brief Title: Stem Cells for the Treatment of Pouchitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decision not to move forward with study.
Sponsor: The Cleveland Clinic (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Amy Lightner, Staff Colorectal Surgeon, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF-Pouchitis
Record Dates: First submitted 2019-11-01; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Pouchitis; Crohn's Disease; Ulcerative Colitis Chronic; Inflammatory Bowel Diseases; Pouch, Ileal
Keywords: Mesenchymal Stem Cells; Crohn's Disease; Inflammatory Bowel Diseases; Pouchitis; Ulcerative Colitis
MeSH Terms: conditions — Pouchitis; Crohn Disease; Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Submucosal endoscopic injection of 60 million allogeneic bone marrow derived mesenchymal stem cells (MSCs) into ileal pouch at baseline and possibly again after 3 months if not completely healed.
  Interventions: Drug: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Drug: Mesenchymal Stem Cells (MSCs) — Endoscopic injection of allogeneic bone marrow derived mesenchymal stem cells (MSCs) to the ileal pouch.
  Other Names: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells (MSCs)

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using allogeneic bone marrow derived mesenchymal stem cells (MSCs) to treat people with medically refractory Pouchitis.

DETAILED DESCRIPTION:
Proctocolectomy with ileal pouch anal anastomosis (IPAA) remains the procedure of choice for patients with chronic ulcerative colitis (CUC). IPAA allows at-risk tissue to be removed with restoration of intestinal continuity while maintaining favorable long-term functional outcomes and quality of life.

While less than 30% of patients experience short-term postoperative morbidity following IPAA, up to 15% of pouches will ultimately fail due to technical or inflammatory complications, the majority of which manifest as a fistula from the pouch to the perianal or vaginal locations. After anastomotic leak, the second leading cause of pouch fistulas is the development of Crohn's disease of the pouch. While the majority of pouches are constructed for CUC, up to 25% will end up having a change in diagnosis to CD which manifests as refractor pouchitis, strictures of the proximal small bowel, or most often as peripouch fistulas. Pouch failure due to refractory pouchitis are notoriously difficult to treat, and reconstructive pouch surgery or transanal repairs are often not offered due to suspicion of recurrent pouchitis following pouch reconstruction. The reality is that patients with refractory pouchitis will end up with a major reconstructive transabdominal operation in a select few for attempt at pouch salvage, or, most likely, a permanent end ileostomy after pouch excision. This can be a devastating outcome in some patients as it impacts body image and quality of life.

Similar to refractory pouchitis, Crohn's related perianal and rectovaginal fistula are other phenotypes of inflammatory bowel disease that are also notoriously difficult to treat with conventional medical and surgical options. Despite an ever expanding repertoire of biologic therapy and surgical intervention, sustained healing rates are less than 30%. This has driven investigators to search for alternative approaches, and in 2003 investigators reported successful healing of a refractory Crohn's rectovaginal fistula following injection of mesenchymal stem cells (MSCs). Following this success, several phase I, II, and III trials designed to study the safety and efficacy of MSCs for perianal CD, all of which have reported encouraging results with superior efficacy compared to conventional medical and surgical therapies. Over 300 perianal CD patients have now been treated without increase in adverse events and no risk of incontinence.

Given the high safety profile, and substantial success in treating perianal CD, the investigators are using a GMP grade allogeneic adipose derived MSCs to establish safety and secondarily monitor for healing in patients with medically refractory pouchitis. This trial will use allogeneic bone marrow derived mesenchymal stem cells (MSCs) to produce regenerative signals which alter the ileal pouch microbiome and local inflammatory mileau. Patients with CD of the pouch suffer chronic immunosuppression and surgical intervention and desperately need an improved therapeutic. The research aims to address the root cause of this inflammation, especially the interactions of the intestinal microbiome and host immune response through a novel therapeutic approach. The specific rationale for MSCs in medical refractory pouchitis is based opon 1) their anti-inflammatory properties; 2) published experience of MSC in this condition and perianal Crohn's fistula demonstrating efficacy and safety; 3) existence of cGMP methods for their isolation and growth.

The study will enroll adult patients with medically refractory pouchitis, whose next option in the treatment plan would be major reconstructive abdominal surgery or pouch excision with a permanent end ileostomy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-75 years of age
2. Residents of the United States
3. Medically refractory pouchitis defined as lack of response to antibiotics, immunomodulators, and/or biologics
4. Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, anti-TNF therapy, anti-integrin and anti-interleukin are permitted if have been on them for at least 2 months prior to study enrollment without change
5. No malignant or premalignant intestinal condition, ruled out on colonoscopy within 90 days of MSC delivery
6. Ability to comply with protocol
7. Competent and able to provide written informed consent
8. Must have failed or have a contraindication to standard medical therapy including anti-TNF, anti-interleukin, or anti-integrin agent

Exclusion Criteria:

1. Inability to give informed consent
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient
3. Specific exclusions:

   * HIV
   * Hepatitis B or C
   * Abnormal CBC at screening
   * Abnormal AST or ALT at screening
4. History of cancer including melanoma (with the exception of localized skin cancers) within 5 years of study enrollment
5. Investigational drug use within thirty (30) days of baseline
6. Pregnant or breastfeeding
7. Multifocal proximal small bowel involvement which resembles Crohn's of the small bowel
8. Evidence of pelvic sepsis and pelvic penetrating fistulizing disease
9. Patients with intestinal diversion above the level of the pouch
10. Neoplasia of pouch
11. Change in medical regimen for pouchitis in the two months prior to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Change from Baseline over 12 months after the MSC injection
  Number of adverse events that occur throughout the study.
Healing | Change from Baseline over 12 months after the MSC Injection
  PDAI endoscopic activity less than or equal to 1, Clinical PDAI score less than or equal to 2, and total PDAI less than or equal to 4

SECONDARY OUTCOMES:
Endoscopic Remission | Change from Baseline over 12 months after the MSC Injection
  PDAI endoscopic activity less than or equal to 1 Mayo Endoscopic score less than or equal to 1, defined as the absence of friability or ulceration
Clinical Remission | Change from Baseline over 12 months after the MSC Injection
  Clinical PDAI score less than or equal to 2 MDPAI score less than or equal to 4
Endoscopic Improvement | Change from Baseline over 12 months after the MSC Injection
  Reduction in the endoscopic PDAI score, but still greater than 1 Reduction in the Mayo endoscopic score, but still greater than 1 Reduction in endoscopic MPDAI score by 2 or more points
Clinical Improvement | Change from Baseline over 12 months after the MSC Injection
  Reduction in the clinical PDAI score of 2 or more points Reduction in the Clinical MPDAI score of 2 or more points Decrease in 24-hour stool frequency
Partial Clinical Healing measured with the Pouchitis Disease Activity Index No No response | Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months after MSC injection
  No improvement in the PDAI overall, endoscopic, or clinical scores No decrease in Mayo endoscopic severity score No decrease in 24 hour stool frequency
Partial Clinical Healing | Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months after MSC injection
  Decrease in C-reactive protein serum levels by greater than 50%
Partial Clinical Healing | Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months after MSC injection
  Decreased mucosal ulceration on pouchoscopy
Partial Clinical Healing | Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months after MSC injection
  Improved healing on endoscopic biopsy or surgical pathology as compared to pre-MSC delivery endoscopic biopsies.
Assess for alloimmune response | Baseline, 1 month, 3 month, 12 month after MSC injection
  Measure HLA Class B Antibody Screening

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Cho YB, Lee WY, Park KJ, Kim M, Yoo HW, Yu CS. Autologous adipose tissue-derived stem cells for the treatment of Crohn's fistula: a phase I clinical study. Cell Transplant. 2013;22(2):279-85. doi: 10.3727/096368912X656045. Epub 2012 Sep 21. PMID 23006344
- [Background] Dietz AB, Dozois EJ, Fletcher JG, Butler GW, Radel D, Lightner AL, Dave M, Friton J, Nair A, Camilleri ET, Dudakovic A, van Wijnen AJ, Faubion WA. Autologous Mesenchymal Stem Cells, Applied in a Bioabsorbable Matrix, for Treatment of Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2017 Jul;153(1):59-62.e2. doi: 10.1053/j.gastro.2017.04.001. Epub 2017 Apr 9. PMID 28400193
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Background] Molendijk I, Bonsing BA, Roelofs H, Peeters KC, Wasser MN, Dijkstra G, van der Woude CJ, Duijvestein M, Veenendaal RA, Zwaginga JJ, Verspaget HW, Fibbe WE, van der Meulen-de Jong AE, Hommes DW. Allogeneic Bone Marrow-Derived Mesenchymal Stromal Cells Promote Healing of Refractory Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2015 Oct;149(4):918-27.e6. doi: 10.1053/j.gastro.2015.06.014. Epub 2015 Jun 25. PMID 26116801
- [Background] Cho YB, Park KJ, Yoon SN, Song KH, Kim DS, Jung SH, Kim M, Jeong HY, Yu CS. Long-term results of adipose-derived stem cell therapy for the treatment of Crohn's fistula. Stem Cells Transl Med. 2015 May;4(5):532-7. doi: 10.5966/sctm.2014-0199. Epub 2015 Mar 31. PMID 25829404
- [Background] Lee WY, Park KJ, Cho YB, Yoon SN, Song KH, Kim DS, Jung SH, Kim M, Yoo HW, Kim I, Ha H, Yu CS. Autologous adipose tissue-derived stem cells treatment demonstrated favorable and sustainable therapeutic effect for Crohn's fistula. Stem Cells. 2013 Nov;31(11):2575-81. doi: 10.1002/stem.1357. PMID 23404825
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896
- [Background] Ciccocioppo R, Bernardo ME, Sgarella A, Maccario R, Avanzini MA, Ubezio C, Minelli A, Alvisi C, Vanoli A, Calliada F, Dionigi P, Perotti C, Locatelli F, Corazza GR. Autologous bone marrow-derived mesenchymal stromal cells in the treatment of fistulising Crohn's disease. Gut. 2011 Jun;60(6):788-98. doi: 10.1136/gut.2010.214841. Epub 2011 Jan 21. PMID 21257987
- [Background] de la Portilla F, Alba F, Garcia-Olmo D, Herrerias JM, Gonzalez FX, Galindo A. Expanded allogeneic adipose-derived stem cells (eASCs) for the treatment of complex perianal fistula in Crohn's disease: results from a multicenter phase I/IIa clinical trial. Int J Colorectal Dis. 2013 Mar;28(3):313-23. doi: 10.1007/s00384-012-1581-9. Epub 2012 Sep 29. PMID 23053677